CLINICAL TRIAL: NCT04952909
Title: A Prospective, Multicenter, Non-Randomized, Single-Arm, Open-Label Clinical Study to Demonstrate the Safety and Effectiveness of the ShortCut™ Device (The ShortCut™ Study)
Brief Title: The ShortCut™ Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pi-cardia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S01-CLN-002
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2023-08

CONDITIONS: Risk of Coronary Obstruction Following Transcatheter Aortic Valve Replacement (TAVR) Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ShortCut™ (Experimental)
  Interventions: Device: ShortCut™

INTERVENTIONS:
Device: ShortCut™ — Splitting bioprosthetic aortic valve leaflets

SUMMARY:
A Prospective, Multicenter, Non-Randomized, Single-Arm, Open-Label Clinical Study to Demonstrate the Safety and Effectiveness of the ShortCut™ device for splitting bioprosthetic aortic valve leaflets in patients who are presented for a valve-in-valve (ViV) transcatheter aortic valve replacement (TAVR) procedure for an approved ViV indication, and who are at risk for TAVR-induced coronary artery ostium obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned to undergo a percutaneous valve-in-valve procedure for an approved valve-in-valve indication due to a failed bioprosthetic valve.
* Written informed consent to participate in the study obtained from the subject or subject's legal representative, according to local regulations, prior to initiation of any study mandated procedure.

Exclusion Criteria:

* An excessive aortic valve leaflet Calcium morphology or anatomy not suitable for the use of the ShortCut™ device.
* Coronary, carotid or vertebral artery disease that, in the opinion of the local Heart Team, should be treated; or treatment of such disease ≤ 1 month prior to index procedure.
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) ≤ 6 months prior to index procedure, or severe neurological disability.
* Myocardial infarction (MI) ≤ 6 weeks prior to index procedure.
* Hemodynamic or respiratory instability.
* Left ventricle ejection fraction < 30%.
* Ongoing severe infection, sepsis or endocarditis.
* Renal insufficiency
* Need for emergency surgery for any reason.
* Life expectancy is less than 1 year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (13):
  - Tucson Medical Center, Tucson, Arizona
  - Smidt Heart Institute Cedars-Sinai Medical, Los Angeles, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center / Atrium Health, Charlotte, North Carolina
  - UPMC Pinnacle, Wormleysburg, Pennsylvania
  - Baylor Scott & White, The Heart Hospital Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
- France (3):
  - CHU de Bordeaux (Bordeaux University Hospital), Bordeaux
  - Institute Mutualiste Montsouris, Paris
  - Clinique Pasteur, Toulouse
- Germany (3):
  - German Heart Institute Berlin, Berlin
  - University Hospital Hamburg, Hamburg
  - Leipzig Heart Institute, Leipzig
- Israel (2):
  - Sha'are Tzedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- United Kingdom (2):
  - Royal Sussex County Hospital, Brighton
  - Leeds General Infirmary, Leeds

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 22 clinical sites from January 2022 to September 2023.
Pre-assignment Details: 66 subjects were found eligible per protocol. 60 subjects were treated with the device (started), after 6 subjects dropped out prior to treatment.
Period: Overall Study
Arm/Group | ShortCut™
Started | 60
30 Days Follow up | 58
90 Days Follow up | 57
Completed | 57
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Includes all patients that were treated with the ShortCut device
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 0
  Unknown or Not Reported | 16
Surgical risk [Count of Participants; unit: Participants]
  Extremely high | 6
  HIgh | 54
Coronary artery disease [Count of Participants; unit: Participants] | 26
Renal impairment [Count of Participants; unit: Participants]
  Severe | 20
  Moderate | 24
  None/mild | 16
Prior coronary artery bypass grafting [Count of Participants; unit: Participants] | 13
Prior stroke [Count of Participants; unit: Participants] | 7
Failed Valve Type [Count of Participants; unit: Participants]
  Surgical Aortic Valve Replacement (SAVR) | 58
  Transcatheter Aortic Valve Replacement (TAVR) | 2
Aortic valve disease [Count of Participants; unit: Participants]
  Aortic Stenosis (AS) | 35
  Aortic Regurgitation (AR) | 7
  Mixed failure (both Aortic Stenosis and Aortic Regurgitation) | 18

OUTCOME MEASURES:

1. Primary Outcome: (Number of Patients With) ShortCut™ Device- and/or ShortCut™ Procedure-related Mortality and All Cause Stroke
Time Frame: Discharge or at 7 days post-procedure, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants
  All-cause mortality | 0
  All-cause stroke | 1
  No ShortCut™ device- and/or ShortCut™ procedure-related mortality and all cause stroke | 59

2. Primary Outcome: (Number of Patients With) Leaflet Splitting Success Using the ShortCut™ Device
Description: Assessed by echo and/or angiography
Time Frame: Intra-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 60

3. Secondary Outcome: (Number of Patients With) All-cause Mortality
Description: (VARC-3) The Valve Academic Research Consortium (VARC) is intended to (i) identify appropriate clinical endpoints and (ii) standardize definitions of these endpoints for transcatheter and surgical aortic valve clinical trials.
  VARC-3 provides an update of the most appropriate clinical endpoint definitions to be used in the conduct of transcatheter and surgical aortic valve clinical research.
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants
  All-cause mortality | 2
  Cardiovascular mortality | 0
  No all-cause mortality | 58

4. Secondary Outcome: (Number of Patients With) All-cause Stroke
Description: as for outcome 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants
  Fatal stroke | 0
  Stroke with disability | 1
  Stroke without disability | 0
  No all-cause stroke | 59

5. Secondary Outcome: (Number of Patients With) Coronary Obstruction
Description: as for outcome 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 3

6. Secondary Outcome: (Number of Patients With) Myocardial Infarction With New Evidence of Coronary Artery Obstruction Requiring Intervention
Description: as for outcome 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 2

7. Secondary Outcome: (Number of Patients With) Major Vascular Complications
Description: as for outcome 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 0

8. Secondary Outcome: (Number of Patients With) Cardiac Tamponade
Description: as for outcome 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 1

9. Secondary Outcome: (Number of Patients With) Acute Kidney Injury
Description: (Acute kidney injury stage 3-4 per VARC-3)
  The Valve Academic Research Consortium (VARC) is intended to (i) identify appropriate clinical endpoints and (ii) standardize definitions of these endpoints for transcatheter and surgical aortic valve clinical trials. VARC-3 provides an update of the most appropriate clinical endpoint definitions to be used in the conduct of transcatheter and surgical aortic valve clinical research.
  * Acute kidney injury stage 3:
    * Increase in serum creatinine >300% (>3.0 X increase) within 7 days compared with baseline
    * Serum creatinine ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of ≥0.5 mg/dL (≥44 mmol/L)
  * Acute kidney injury stage 4:
    * AKI requiring new temporary or permanent renal replacement therapy
  No differentiation was made between the stages when assessing the outcome.
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 2

10. Secondary Outcome: (Number of Patients With) Access-related Type 3-4 Bleeding
Description: (VARC-3) The Valve Academic Research Consortium (VARC) is intended to (i) identify appropriate clinical endpoints and (ii) standardize definitions of these endpoints for transcatheter and surgical aortic valve clinical trials. VARC-3 provides an update of the most appropriate clinical endpoint definitions to be used in the conduct of transcatheter and surgical aortic valve clinical research.
  * Type 3 bleeding:
    * Overt bleeding causing hypovolemic shock or severe hypotension (systolic blood pressure <90 mmHg lasting >30 min and not responding to volume resuscitation) or requiring vasopressors or surgery (BARC 3b)
    * Overt bleeding requiring reoperation, surgical exploration, or reintervention for the purpose of controlling bleeding (BARC 3b, BARC 4)
    * Overt bleeding requiring a transfusion of ≥5 units of whole blood/red blood cells (BARC 3a)
    * Overt bleeding associated with a hemoglobin drop ≥5 g/dL (≥3.1 mmol/L) (BARC 3b)
  * Type 4 bleeding:
    * Overt bleeding leading
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 0

11. Secondary Outcome: (Number of Patients With) Freedom From Coronary Artery Ostia Obstruction Related to the Intervened Leaflet
Time Frame: 30 days post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 57

12. Secondary Outcome: (Number of Patients With) Freedom From Coronary Artery Intervention Related to the Intervened Leaflet
Time Frame: 30 days post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 56

13. Secondary Outcome: (Number of Patients With) ShortCut™ Technical Success
Description: Technical success is defined as a composite of the following:
  * Successful access, delivery, and retrieval of the ShortCut™ device
  * Freedom from ShortCut™ device- and/or ShortCut™ procedure-related mortality
  * Freedom from ShortCut™ device- and/or ShortCut™ procedure-related: Surgery or intervention, Major vascular or access-related complications, Cardiac structural complication.
Time Frame: At exit from procedure room
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 59

14. Other Pre Specified Outcome: (Number of Patients With) All-cause Mortality
Description: as for outcome 3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 3

15. Other Pre Specified Outcome: (Number of Patients With) Stroke
Description: as for outcome 3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 1

16. Other Pre Specified Outcome: (Number of Patients With) Myocardial Infarction With New Evidence of Coronary Artery Obstruction Requiring Intervention
Description: as for outcome 3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ShortCut™
Number analyzed (Participants) | 60
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported from point of index procedure until 90 days post procedure
Arm/Group | ShortCut™
All-Cause Mortality (participants affected / at risk) | 3/60
Serious Adverse Events (participants affected / at risk) | 13/60
Other Adverse Events (participants affected / at risk) | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShortCut™ (N=60)
All-cause stroke (Nervous system disorders) | 1 (1) — Per VARC-3
Coronary obstruction (Cardiac disorders) | 3 (3) — Per VARC-3
Myocardial Infarction with new evidence of coronary artery obstruction requiring intervention (Cardiac disorders) | 2 (2) — Per VARC-3
Cardiac tamponade (Cardiac disorders) | 1 (1) — Per VARC-3
Acute kidney injury stage 3-4 (Renal and urinary disorders) | 2 (2) — Per VARC-3
Permanent pacemaker (Cardiac disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShortCut™ (N=60)
Left Bundle Branch Block (LBBB) (Cardiac disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT04952909/Prot_SAP_000.pdf